CLINICAL TRIAL: NCT01492231
Title: The Clinical Impact and Outcomes of Interventional Endoscopy Procedures
Status: Enrolling by invitation | Type: Observational
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Kenneth J. Chang, Professor of Clinical Medicine, University of California, Irvine
Other Study IDs: 20086258
Record Dates: First submitted 2011-12-02; First posted 2011-12-14 (Estimated); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Gastrointestinal Diseases
Keywords: gastroenterology; Endoscopy, Digestive System; Endosonography; Endoscopic Retrograde Cholangiopancreatography; gastrointestinal endoscopy
MeSH Terms: conditions — Gastrointestinal Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Chart Review: Chart review of patients who had a procedure done at H. H. Chao Comprehensive Digestive Disease Center

SUMMARY:
The main purpose of the protocol is to collect and evaluate performance data after patients undergoing various interventional endoscopy procedures performed at H. H. Chao Comprehensive Digestive Disease Center (CDDC).

DETAILED DESCRIPTION:
In general, the outcome data includes clinical management, hospitalization, and complications; to determine costs associated with endoscopy procedures; to determine performance data including technical success, procedure time, rate of repeat interventions; to compare endoscopy performance and outcome data collected at University of California, Irvine (UCI) and results from other institutions previously published in the literature. Additional parameters might be collected for specific interventional endoscopy procedures.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are 18 years of age or older
* Subjects who are scheduled for a procedure at the H. H. Chao Comprehensive Digestive Disease Center (CDDC).

Exclusion Criteria:

* Subjects who are not 18 years of age or older
* Subjects who are scheduled for a procedure at the H. H. Chao Comprehensive Digestive Disease Center (CDDC).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with gastrointestinal disease(s) undergoing various interventional endoscopy procedures performed at H. H. Chao Comprehensive Digestive Disease Center (CDDC).
Sampling Method: Probability Sample
Enrollment: 3500 (Estimated)
Dates: Start 2008-11; Primary Completion 2025-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Collect and clinical management data | Day of procedure up to 5 years for follow-up (if needed).
  Outcome data includes clinical management (such as hospitalization information, and complications, costs associated with endoscopy procedures, etc.).

SECONDARY OUTCOMES:
Collect Performance Data | Day of procedure up to 5 years for follow-up (if needed).
  Outcome performance data (such as, technical success, procedure time, rate of repeat interventions, lab/pathology results, etc.)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Chang, MD, Principal Investigator — University of California, Irvine
Locations (1):
- H. H. Chao Comprehensive Digestive Disease Center, Orange, California, United States